CLINICAL TRIAL: NCT00398073
Title: Injection of AJCC Stage IIB, IIC, III and IV Melanoma Patients With Mouse gp100 DNA: A Pilot Study to Compare Intramuscular Jet Injection With Particle Mediated Delivery
Brief Title: Vaccine Therapy in Treating Patients With Stage IIB, Stage IIC, Stage III, or Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-113; MSKCC-06113
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma; ciliary body and choroid melanoma, medium/large size; ciliary body and choroid melanoma, small size; recurrent intraocular melanoma; metastatic intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Injections, Intramuscular

ARMS (2):
- mouse gp100 DNA via PMED (Experimental): patients will be randomized to mouse gp100 DNA delivered via gold particles using the PowderMed delivery system (ND10, described above). Two actuations/day will be administered every two weeks for 4 months for a total of 16 actuations. Each actuation consists of 2 μg of plasmid DNA coated onto 1000 μg of gold. The total dose of plasmid DNA given will be 32 μg DNA on 16,000 μg gold.
  Interventions: Biological: mouse gp100 plasmid DNA vaccine; Device: The Dermal PowderMed® devices
- mouse gp100 DNA injections intramuscularly (Experimental): patients will be injected with 1000 μg of mouse gp100 plasmid DNA intramuscularly. Two injections/day will be administered every two weeks for 4 months (4000 ug of mouse gp100 plasmid/month) for 16 vaccinations.
  Interventions: Biological: mouse gp100 plasmid DNA vaccine; Other: intramuscularly (IM injection)

INTERVENTIONS:
Biological: mouse gp100 plasmid DNA vaccine
Device: The Dermal PowderMed® devices
  Arms: mouse gp100 DNA via PMED
Other: intramuscularly (IM injection)
  Arms: mouse gp100 DNA injections intramuscularly

SUMMARY:
RATIONALE: Vaccines made from DNA may help the body build an effective immune response to kill tumor cells. Giving the vaccine in different ways may make a stronger immune response and kill more tumor cells.

PURPOSE: This randomized clinical trial is studying two different ways of giving vaccine therapy to compare how well they work in treating patients with stage IIB, stage IIC, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and feasibility of particle-mediated epidermal delivery (PMED) immunization comprising mouse gp100 plasmid DNA vaccine in patients with stage IIB, IIC, III, or IV melanoma.
* Compare the immunologic response induced with PMED vs intramuscular jet injection methods of vaccination in these patients.

Secondary

* Observe patients with measurable tumor for evidence of any antitumor response generated after vaccination.
* Assess for disease relapse in patients treated with this vaccine.

OUTLINE: This is a randomized, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive mouse gp100 plasmid DNA vaccine by particle-mediated epidermal delivery on days 1, 3, 5, 8, 22, 24, 26, 29, 43, 45, 47, 50, 64, 66, 68, and 71.
* Arm II: Patients receive mouse gp100 plasmid DNA vaccine by intramuscular jet injection on days 1, 3, 5, 8, 22, 24, 26, 29, 43, 45, 47, 50, 64, 66, 68, and 71.

After completion of study treatment, patients are followed periodically for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Stage IIB, IIC, III, or IV disease

    * Patients free of disease after surgical resection must meet 1 of the following criteria:

      * Refused high-dose interferon alfa
      * Recurrence while on interferon alfa
    * Patients with stage IIB, IIC, or III disease must have already undergone initial standard therapy (i.e., surgery) for the disease
* Choroidal (uveal) melanoma allowed provided 1 of the following criteria is met:

  * Basal diameter > 16 mm
  * Basal height > 8 mm
  * Involvement of the ciliary body with tumor
* HLA-A*0201 positive
* Negative serum antidouble-stranded DNA antibody screen
* No known brain metastases

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* WBC ≥ 3,000/mm^3
* Lactic dehydrogenase ≤ 2 times upper limit of normal (ULN)
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.5 times ULN
* Albumin ≥ 3.5 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Weight ≥ 25 kg
* No preexisting choroidal eye disease
* No serious underlying medical conditions that could be exacerbated by study participation (i.e., active infections requiring antimicrobial drugs or active bleeding)
* No allergy to gold (i.e., gold jewelry)
* No evidence of any condition at the proposed site(s) of vaccine administration that might interfere with the interpretation of local skin reactions, including any of the following:

  * Damaged skin
  * Moles
  * Scars
  * Tattoos
  * Marks
* No prior medical condition or use of medication (e.g., corticosteroids) that might make it difficult for the patient to complete the full course of treatment or to respond immunologically to vaccines
* No history or evidence (within the past 5 years) of a physician-diagnosed chronic or recurrent inflammatory skin disease at the proposed site of vaccine administration, including any of the following:

  * Psoriasis
  * Eczema
  * Atopic dermatitis
  * Hypersensitivity
* No history of keloid formation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy, immunotherapy, or radiotherapy (6 weeks for nitrosoureas) and recovered
* No prior immunization with any class of vaccine containing gp100 peptide
* No other concurrent investigational agents
* No other concurrent systemic therapy or radiotherapy

Ages: 1 Year to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jedd D. Wolchok, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 1_Particle-medicated Epidermal Delivery Group (Gene Gun): patients will be randomized to mouse gp100 DNA delivered via gold particles using the PowderMed delivery system (ND10, described above). Two actuations/day will be administered every two weeks for 4 months for a total of 16 actuations. Each actuation consists of 2 μg of plasmid DNA coated onto 1000 μg of gold. The total dose of plasmid DNA given will be 32 μg DNA on 16,000 μg gold.
  mouse gp100 plasmid DNA vaccine
- 2_IM Injection (Bioinjector): patients will be injected with 1000 μg of mouse gp100 plasmid DNA intramuscularly. Two injections/day will be administered every two weeks for 4 months (4000 ug of mouse gp100 plasmid/month) for 16 vaccinations.
  mouse gp100 plasmid DNA vaccine
Period: Overall Study
Arm/Group | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) | 2_IM Injection (Bioinjector)
Started | 18 | 17
Completed | 17 | 17
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) | 2_IM Injection (Bioinjector) | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 8
  Male | 15 | 11 | 26
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Evulated for Toxicity and Safety
Description: All toxicity will be graded according to the National Cancer Institute (NCI) Common Toxicity Criteria v3.0.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) | 2_IM Injection (Bioinjector)
Number analyzed (Participants) | 17 | 17
participants | 17 | 17

2. Primary Outcome: Number of Participants With a T-cell Response
Description: T-cell response: Peripheral blood lymphocytes will be tested for reactivity against gp100 using an IFN-y ELISPOT, intracellular cytokine staining or MHC tetramer assay. If T-cell reactivity is induced, additional samples may be drawn to determine the duration of this reactivity. Follow-up blood samples require only 20-30 ml. MHC tetramer assays and intracellular flow cytometry studies may also be performed.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) | 2_IM Injection (Bioinjector)
Number analyzed (Participants) | 17 | 17
participants | 17 | 17

3. Secondary Outcome: Number of Participants With Response
Description: In patients with measurable disease, the RECIST criteria for anti-tumor effect will be used. Lesions will be defined as measurable if they can be accurately measured in at least one dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm by spiral CT scan.Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) | 2_IM Injection (Bioinjector)
Number analyzed (Participants) | 17 | 17
participants | 17 | 17

ADVERSE EVENTS:
Arm/Group | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) | 2_IM Injection (Bioinjector)
Serious Adverse Events (participants affected / at risk) | 3/17 | 1/17
Other Adverse Events (participants affected / at risk) | 5/17 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) (N=17) | 2_IM Injection (Bioinjector) (N=17)
Allergy/Immunology, other (Immune system disorders) | 1 (1) | 0 (0)
Allergy/Immunology, other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Edema: limb (Blood and lymphatic system disorders) | 1 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1_Particle-medicated Epidermal Delivery Group (Gene Gun) (N=17) | 2_IM Injection (Bioinjector) (N=17)
AST, SGOT (Metabolism and nutrition disorders) | 1 | 0
Bilirubin (hyperbilirubinemia) (Hepatobiliary disorders) | 2 | 3
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 3 | 3
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes